CLINICAL TRIAL: NCT05644613
Title: Effect Of Aerobic Exercises On Land Versus Aerobic Exercises In Water In The Management Of Premenstrual Syndrome In Adolescent Girls
Brief Title: Comparative Study Between The Effect Of Aerobic Exercises On Land and Aerobic Exercises In Water On PMS Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mariam Hossam El Ebrashy (Other)
Responsible Party: Sponsor-Investigator, Mariam Hossam El Ebrashy, Lectruer, Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Premenstrual Syndrome
Keywords: premenstrual syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Exercise; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Active Comparator): will consist of (20) adolescent girls age ranged from 14-17 suffering from PMS without any pathological cause they will receive an aerobic exercise on land in form of walking on the treadmill for 20 min 3 times per week for 3 months.
  Interventions: Other: aerobic exercise on land
- GROUP B (Active Comparator): will consist of (20) adolescent girls age ranged from 14-17 suffering from PMS without any pathological cause they will receive an aerobic exercises in water in form of walking on the treadmill for 20 min 3 times per week for 3 months
  Interventions: Other: aerobic exercise in water

INTERVENTIONS:
Other: aerobic exercise on land — aerobic exercise on land in form of walking on the treadmill
  Arms: GROUP A
Other: aerobic exercise in water — aerobic exercises in water in form of walking on the treadmill
  Arms: GROUP B

SUMMARY:
Many girls experience premenstrual syndrome PMS which is re a group of physical, cognitive, affective, and behavioural symptoms that occur cyclically during the luteal phase of the menstrual cycle and resolve at or within a few days of the onset of menstruation. In young adolescents symptoms might particularly affect school functions, and social interactions in a negative ways in this study we will figure out the effect of 2 kinds of exercises in the management of this syndrome.

DETAILED DESCRIPTION:
Fourty adolescent girls were divided randomly into two equal groups, Group (A) will consist of (20) adolescent girls age ranged from 14-17 suffering from PMS without any pathological cause they will receive an aerobic exercise on land in form of walking on the treadmill for 20 min 3 times per week for 3 months. Group (B) will consist of (20) adolescent girls age ranged from 14-17 suffering from PMS without any pathological cause they will receive an aerobic exercises in water in form of walking on the treadmill for 20 min 3 times per week for 3 months the assessment of the PMS symptoms will be done by Premenstrual distress questionnaire

ELIGIBILITY:
Inclusion Criteria:

* All participants virgin females.
* Their age ranged from 14 to 17 years old
* their body mass index (BMI) ≥ 18 ≤ 25 kg/m2.
* They are clinically and medically stable during the study,
* they have regular menstrual cycle of 23 to 35 days and not participated any type of unusual diet during the period of the study.

Exclusion Criteria:

* All females in this study are free from: cardiopulmonary or orthopaedic problems, taking any hormonal drugs for three months at least, participating in any form of activity rather than the prescribed one in the study, any abnormality in ovulation or pelvic inflammatory diseases (PID).

Ages: 14 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-03-02 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Premenstrual syndrome symptoms | 3 months
  PREMENSTRUAL SYNDROME QUESTIONNAIRE

CONTACTS AND LOCATIONS:
Overall Officials: Mina Atef, Phd, Study Director — Badr University
Locations (1):
- Badr University, Cairo, Egypt